CLINICAL TRIAL: NCT03650374
Title: Effects of Contralateral Strength Training on Postoperative Strength Deficits in the Immobilized Lower Extremity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01100
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Meniscus; Detachment, Current Injury
Keywords: Meniscus root tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): standard of care postoperative rehabilitation.
  Interventions: Other: Standard of Care Rehabilitation
- Group 2 (Experimental): experimental strength training
  Interventions: Other: Experimental Strength Training

INTERVENTIONS:
Other: Standard of Care Rehabilitation — Knee flexion and extension strength training exercises for the contralateral (non-operative) lower extremity in addition to standard of care postoperative rehabilitation.
  Arms: Group 1
Other: Experimental Strength Training — Will be performed with moderate resistance and will require moderate effort. Exercises will include unilateral leg presses, lunges, step ups, and step downs. These exercises are performed as standard of care but are not typically introduced into the physical therapy regimen until 10-12 weeks postoperatively. In the experimental group, these exercises will be introduced starting with the first postoperative physical therapy session, but only for the contralateral (non-operative) leg.
  Arms: Group 2

SUMMARY:
This is a prospective, randomized controlled trial that will enroll patients undergoing unilateral meniscal root repair or meniscus transplant. The objective of this study is to determine if immediate postoperative strength training of the contralateral (non-surgical) lower extremity reduces postoperative loss of strength in an immobilized lower extremity.

After the completion of surgery, patients will be randomized to either the experimental treatment (Group 1) or control group (Group II)for postoperative rehabilitation.

DETAILED DESCRIPTION:
Group I will receive knee flexion and extension strength training exercises for the contralateral (non-operative) lower extremity in addition to standard of care postoperative rehabilitation. The experimental strength training will be performed with moderate resistance and will require moderate effort. Exercises will include unilateral leg presses, lunges, step ups, and step downs. These exercises are performed as standard of care but are not typically introduced into the physical therapy regimen until 10-12 weeks postoperatively. In the experimental group, these exercises will be introduced starting with the first postoperative physical therapy session, but only for the contralateral (non-operative) leg.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for meniscal root repair
* Patient is indicated for meniscus transplant
* Patient is at least 18 years of age
* Patient is expected to survive at least 1 year beyond surgery
* Patient has intact lower extremities bilaterally
* Patient is willing to participate by complying with pre-and post-operative visit requirements
* Patient is willing and able to review and sign a study informed consent form

Exclusion Criteria:

* Lower extremity musculoskeletal defects
* Systemic neuromuscular disorders
* Failure to complete pre-operative BIDOEX strength assessment
* Failure to complete pre-operative self-assessment score intake forms

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
KOOS | 6 Weeks, 3 Months, 6 Months
  A patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
PI (Dr. Lomas) will be the only individual viewing and handling IPD